CLINICAL TRIAL: NCT02674243
Title: Efficacy of Iodopovidone Versus Talc in Palliative Malignant Pleural Effusion: a Randomized Controlled Trial Study
Brief Title: Efficacy of Iodopovidone Versus Talc in Palliative Malignant Pleural Effusion
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Apichat Tantraworasin, Assistant Professor, Chiang Mai University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 03315
Record Dates: First submitted 2016-02-01; First posted 2016-02-04 (Estimated); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Malignant Pleural Effusion
Keywords: Malignant pleural effusion; Pleurodesis; Talc; Iodopovidone solution; Povidone-iodine
MeSH Terms: conditions — Pleural Effusion, Malignant | interventions — Povidone-Iodine; Talc

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Iodopovidone group (Experimental): Patients who will be randomized for using iodopovidone solution for pleurodesis.
  Interventions: Drug: Iodopovidone solution
- Talc group (Active Comparator): Patients who will be randomized for using Talc for pleurodesis.
  Interventions: Drug: Talc

INTERVENTIONS:
Drug: Iodopovidone solution — In this group, iodopovidone solution will be used as pleurodesis substance
  Other Names: povidone-iodine solution
  Arms: Iodopovidone group
Drug: Talc — In this group, Talc will be used as pleurodesis substance
  Other Names: Talcum powder
  Arms: Talc group

SUMMARY:
This is prospective randomized control trial study. The aim of this study is to evaluate the efficacy of Iodopovidone solution for pleurodesis in palliative malignant pleural effusion (MPE) patients comparing to Talc. All adult patients who diagnosed MPE by cytology regardless primary tumor between December 1, 2015 and November 29, 2016 at Maharaj Nakorn Chiang Mai Hospital, Chiang Mai University, Chiang Mai, Thailand will be enrolled in this study. The inform and consent will be applied in all patients before treatment. Patients will be randomized to two groups; Iodopovidone group (intervention group) and Talc group (control group)

DETAILED DESCRIPTION:
Background and Rationale: Malignant pleural effusion (MPE) defined as presenting malignant cell in pleural effusion. It is usually found in advanced stage cancer or cancer of pleura. Most common primary tumor causing MPE is lung cancer (37%) followed with breast cancer (16%). From previous studies, when MPE was diagnosed, the median survival was only 3-12 months depending on primary tumor. In lung cancer, median survival for stage IV with MPE was only 4 months. However, quality of life of patient is also important. These patients should have less suffer from MPE. In recent era, chemotherapy, targeted therapy and immunotherapy are very useful for advanced stage cancer patients. They can prolong survival in such patients. Therefore, pleurodesis had role for palliative treatment hoping these patient have better quality of life. Talc (composed of oxygen, silicate, magnesium and carbon) has been used as one of common substances for chemical pleurodesis since 1935 by Norman Bethune with high efficacy (90%). However, it can cause a serious complication such as acute respiratory distress syndrome (ARDS). Although an incidence of ARDS is not too high, it can make patients died, therefore, other substances have been studied instead of using Talc. Iodopovidone has been one of interesting substances used as pleurodesis substance since 2006. It is low cost, and available. One meta-analysis of 13 observational studies with 499 patients found that iodopovidone was safe with success rate of pleurodesis was 70-100%. The most common side effect was chest pain. Previously, only two randomized control trial studies reported the efficacy of iodopovidone solution comparing to Talc for pleurodesis. They found that there were no statistical significant difference either efficacy or safety between two substances. The limitation of those studies is small sample size, therefore, we would like to compare the efficacy of iodopovidone solution for chemical pleurodesis with Talc.

Objectives: To compare the efficacy of Iodopovidone solution with Talc for pleurodesis in MPE Research methodology: This is a prospective randomized control trial. All adult patients who diagnosed MPE by cytology regardless primary tumor between December 1, 2015 and November 29, 2016 at Maharaj Nakorn Chiang Mai Hospital, Chiang Mai University, Chiang Mai, Thailand will be enrolled in this study. Patients will be randomized to two groups; Iodopovidone group (intervention group) and Talc group (control group). The efficacy of both groups will be compared.

ELIGIBILITY:
Inclusion Criteria:

1. All MPE proved by cytology
2. After pleural effusion was released by chest tube drainage, lung was fully expanded

Exclusion Criteria:

1. Patients who have Karnofsky performance state ≤ 40
2. History of iodine allergy
3. History of morphine allergy
4. Abnormal thyroid hormones.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-11; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Success of treatment | 7 days
  Success of treatment defined as chest drain can be removed within 1 week after intervention

SECONDARY OUTCOMES:
Amount of pleural effusion after pleurodesis | Until chest drain removal, an average of 7 days
  Observing amount of pleural effusion after intervention comparing between both groups
Side effect | with 24 hours after intervention
  Side effects are chest pain, fever, and respiratory failure.
Length of hospital stay | From date of randomization until the date of discharge or date of death from any cause, whichever came first, assessed up to 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Apichat Tantraworasin, Principal Investigator — Chiang Mai University
Locations (1):
- Department of surgery, Faculty of medicine, Chiang Mai University Hospital, Chiang Mai, Chaing Mai, Thailand

IPD SHARING:
Plan to Share IPD: Undecided